CLINICAL TRIAL: NCT06461221
Title: Individualized Focused Ultrasound Stimulation of the Brain to Enhance Alertness and Cognitive Performance
Brief Title: tFUS to Enhance Alertness and Performance
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding terminated prior to initiation.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Attune Neurosciences Inc (Industry); Nano-Bio Materials Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00133395; NBRFP23 P31 (Other Grant/Funding Number: Nano-Bio Materials Consortium)
Record Dates: First submitted 2024-04-19; First posted 2024-06-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Reaction Time; Alertness

STUDY DESIGN:
Intervention Model Description: Each participant receives 4 stimulation conditions in a counterbalanced order across 4 visits (1 stimulation condition/visit)
Who Masked: Participant, Investigator
Masking Description: Double-blind sham-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Focused Ultrasound Dose #1 (Experimental): Focused Ultrasound will be administered using high frequency stimulation as condition 1. Stimulation will last 1-10 minutes.
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound Dose #2 (Experimental): Focused Ultrasound will be administered using medium frequency stimulation as condition 2. Stimulation will last 1-10 minutes.
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound Dose #3 (Experimental): Focused Ultrasound will be administered using low frequency stimulation as condition 4. Stimulation will last 1-10 minutes.
  Interventions: Device: Transcranial Focused Ultrasound
- Focused Ultrasound Dose #4 (Sham Comparator): Focused Ultrasound will be administered using the sham condition.
  Interventions: Device: Transcranial Focused Ultrasound

INTERVENTIONS:
Device: Transcranial Focused Ultrasound — Using MRI-guided targeting, we will administer focused ultrasound in one of the 4 stimulation conditions
  Arms: Focused Ultrasound Dose #1
Device: Transcranial Focused Ultrasound — Using MRI-guided targeting, we will administer focused ultrasound in one of the 4 stimulation conditions
  Arms: Focused Ultrasound Dose #2
Device: Transcranial Focused Ultrasound — Using MRI-guided targeting, we will administer focused ultrasound in one of the 4 stimulation conditions
  Arms: Focused Ultrasound Dose #3
Device: Transcranial Focused Ultrasound — Using MRI-guided targeting, we will administer focused ultrasound in one of the 4 stimulation conditions
  Arms: Focused Ultrasound Dose #4

SUMMARY:
The investigators goal is to target FUS energy to the centromedian nucleus of the thalamus (CMT), the core of arousal, which is inaccessible by traditional non-invasive neuromodulation devices. The CMT is an ideal stimulation target for augmenting alertness, as it is intimately linked with the cortex through the well described thalamocortical circuit to entrain network oscillations.

DETAILED DESCRIPTION:
In this research study, the investigators will utilize a novel wearable device (ATTN201) to test the dose-response effects of FUS stimulation of the centromedian nucleus of the thalamus (CMT) on alertness, cognitive performance, and reaction time, as well as sleep EEG recordings. Unlike existing technologies, the device in this study will use offline MRI guidance, which is not needed during the actual treatment, allowing users for the first time to sleep and comfortably wear the device out of the clinic. This unique offline MRI guidance approach uses the device's precise head registration and brain anatomy to allow for customized and repeatable tFUS delivery to the CMT.

For this study, the investigators will recruit up to 36 healthy subjects for a safety study that will objectively assess brain parenchyma morphology, and neuropsychiatric and neuropsychological function, following tFUS exposure of the CMT. EEG recordings during parametric sweeps will be obtained for observation of changes in brain network activity.

ELIGIBILITY:
Inclusion Criteria:

* 22 - 55 y.o.
* Endorse good health with no history of mental or physical illness
* Negative urine pregnancy test if female
* Willingness to adhere to the FUS study schedule and assessments
* Able to read consent document and provide informed consent.
* English is a first or primary fluent language.

Exclusion Criteria:

* Any current psychiatric diagnosis or current Clinical Global Impression ratings of psychiatric illness > 1
* Neurodevelopmental disorders, history of CNS disease, concussion, overnight hospitalization, or other neurologic sequela, tumors, seizures, meningitis, encephalitis, or abnormal CT or MRI of the brain
* Any psychotropic medication is taken within 5 half-lives of procedure time
* Any head trauma resulting in loss of consciousness
* Visual impairment (except the use of glasses)
* Inability to complete cognitive testing
* Active participation or plan for enrollment in another evidence-based clinical trial affecting the psychosocial function
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) or taking medications including stimulants, modafinil, thyroid medication, or steroids
* Implanted devices/ferrous metal of any kind
* History of seizure or epilepsy, currently taking medications that lower seizure thresholds
* Claustrophobia or other conditions that would prevent the MRI assessment.
* Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term).
* Urine Pregnancy Test: If the subject is a woman of childbearing potential and /or a man capable of fathering a child before, during, and/or after participation precautions should be taken. Examples of acceptable methods of birth control for participants involved in the study include birth control pills, patches, IUDs, condoms, sponges, diaphragm with spermicide, or avoiding sexual activity that could cause the subject to become pregnant.
* Inability to adhere to the treatment schedule.
* Inability to fit the wearable device to the user's head.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
EEG changes pre- to post-FUS | 2 years
  Frequency band analysis of EEG data
Reaction time on Psychomotor vigilance task | 2 years
  Measuring reaction time on PVT pre- to post-FUS

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States